CLINICAL TRIAL: NCT02649738
Title: Use of Preserved Corneal Tissue Inlay to Treat Keratoconus
Brief Title: Corneal Tissue Inlay for Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEI-Tissue-Inlay
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Keratoconus
Keywords: keratoconus; corneal tissue inlay
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Corneal tissue inlay (Experimental): The treated cornea will be implanted with a thin disc of preserved corneal tissue
  Interventions: Procedure: Corneal tissue inlay

INTERVENTIONS:
Procedure: Corneal tissue inlay — A mid-stomal pocket will be made into the cornea with a femtosecond laser (Intralase). A small disc of preserved corneal tissue will then be placed into the pocket

SUMMARY:
This study will evaluate the outcomes of placing preserved corneal tissue within the keratoconic cornea in order to enhance thickness, stability, and optical conformation.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the outcomes of placing preserved corneal tissue within the corneal stroma in keratoconus patients as a means of enhancing thickness, stability, and optical conformation.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age, male or female, of any race
* Provide written informed consent and sign a HIPAA form
* Willingness and ability to follow all instructions and comply with schedule for follow-up visits
* For females: Must not be pregnant
* Having topographic evidence of keratoconus which is graded as moderate or severe keratoconus.

Exclusion Criteria:

* Contraindications, sensitivity or known allergy to the use of the test article(s) or their components
* If female, pregnant
* Eyes classified as either normal, atypical normal, keratoconus suspect or mild keratoconus on the severity grading scheme
* Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications For example: a history of corneal disease (e.g., herpes simplex, herpes zoster keratitis, corneal melt, corneal dystrophy, etc.)
* A history of delayed corneal healing in the eye to be treated
* Have used an investigational drug or device within 30 days of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Corneal tissue inlay for keratoconus | 6 months
  Change in maximum keratometry on corneal topography
Corneal tissue inlay for keratoconus | 6 months
  Uncorrected visual acuity
Corneal tissue inlay for keratoconus | 6 months
  Best spectacle corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, MD, Principal Investigator — Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institue - Hersh Vision Group, Teaneck, New Jersey, United States

REFERENCES:
- [Derived] Greenstein SA, Yu AS, Gelles JD, Eshraghi H, Hersh PS. Corneal tissue addition keratoplasty: new intrastromal inlay procedure for keratoconus using femtosecond laser-shaped preserved corneal tissue. J Cataract Refract Surg. 2023 Jul 1;49(7):740-746. doi: 10.1097/j.jcrs.0000000000001187. PMID 36943309